CLINICAL TRIAL: NCT03314389
Title: The Corneal and Conjunctiva Sensation Before and After Pterygium Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ofira Zloto, Principal Investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SHEBA-17-4417-OZ-CTIL
Record Dates: First submitted 2017-10-09; First posted 2017-10-19 (Actual); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Pterygium
Keywords: Cochet bonnet esthesiometer
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cochet bonnet esthesiometer (Experimental): To examine sensation
  Interventions: Device: Cochet bonnet esthesiometer

INTERVENTIONS:
Device: Cochet bonnet esthesiometer — Cochet bonnet esthesiometer- To examine sensation

SUMMARY:
The purpose of this current study is to examine the sensation of the corneal and conjunctiva sensation before and after pterygium surgeries by Cochet bonnet esthesiometer and to examine epidemiological, clinical and imaging factors the influence the sensation

ELIGIBILITY:
Inclusion Criteria:

* Patients that suppose to undergo pterigyum surgery

Exclusion Criteria:

* Patients with anterior segment diseases Patients that underwent anterior segment surgeries Patients with 7th nerve palsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
To sensation before and after pterygium surgeries as measured by Cochet bonnet esthesiometer | Before surgery compare to one week+ one month+three months after surgery
  The change in sensation in the cornea and conjunctiva after pterygium surgery as measured by Cochet bonnet esthesiometer

SECONDARY OUTCOMES:
To examine the change in dry eye syndrome that may predicate the change in sensation after pterygium surgery | Before surgery compare to one week+ one month+three months after surgery
  Dry eye will be measured by Tear break up time
To examine the change in dry eye syndrome that may predicate the change in sensation after pterygium surgery | Before surgery compare to one week+ one month+three months after surgery
  Dry eye will be measured by Schrimer test
To examine the change in dry eye syndrome that may predicate the change in sensation after pterygium surgery | Before surgery compare to one week+ one month+three months after surgery
  Dry eye will be measured by lissamine green test
To examine the change in visual acuity that may predicate the change in sensation after pterygium surgery | Before surgery compare to one week+ one month+three months after surgery
  Visual acuity will be measured by Snellen chart
To examine the change in refraction that may predicate the change in sensation after pterygium surgery: | Before surgery compare to one week+ one month+three months after surgery
  Refraction will be measured by autorefractometer
To examine the change in anterior chamber that may predicate the change in sensation after pterygium surgery: | Before surgery compare to one week+ one month+three months after surgery
  Anterior chamber slit lamp examination
To examine the change in imaging of anterior segment that may predicate the change in sensation after pterygium surgery: | Before surgery compare to one week+ one month+three months after surgery
  Anterior Chamber Optical coherence tomography( AC-OCT)
To examine the Recurrence of pterygium | one week+ one month+three months after surgery
  Recurrence of pterygium as examined in slit lamp examination

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sakarya Y, Sakarya R, Kara S. Reversal of sensation of conjunctival autograft after pterygium surgery. Eur J Ophthalmol. 2012;22 Suppl 7:S11-6. doi: 10.5301/ejo.5000082. PMID 22081668
- [Result] Julio G, Campos P, Pujol P, Munguia A, Mas-Aixala E. Determining Factors for Fast Corneal Sensitivity Recovery After Pterygium Excision. Cornea. 2016 Dec;35(12):1594-1599. doi: 10.1097/ICO.0000000000000932. PMID 27362880
- [Result] Pujol P, Julio G, Barbany M, Asaad M. Healing indicators after pterygium excision by optical coherence tomography. Ophthalmic Physiol Opt. 2015 May;35(3):308-14. doi: 10.1111/opo.12206. Epub 2015 Mar 31. PMID 25833130